CLINICAL TRIAL: NCT00325481
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of a Bivalent Vaccine of New 6:2 Influenza Virus Reassortants in Healthy Adults
Brief Title: Study To Evaluate the Safety of Bivalent Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP134
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist

INTERVENTIONS:
Drug: FluMist

SUMMARY:
To assess the safety of a bivalent vaccine of two new influenza virus reassortants in healthy adults prior to the release of the trivalent vaccine (FluMist) containing them.

DETAILED DESCRIPTION:
This prospective, randomized, double blind, placebo-controlled release study will enroll approximately 300 healthy adults 18-49 years of age. Eligible subjects will be randomly assigned in a 4:1 fashion to receive a single dose of bivalent vaccine or placebo by intranasal spray. This study will be conducted at multiple sites in the United States. Randomization will be stratified by site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 49 years of age (not yet reached their 50th birthday) at the time of study vaccination
* Healthy by medical history and health assessment
* Sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral, implanted, injectable, or transdermal contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for at least 30 days prior to study vaccination, and must agree to continue using such precautions for at least 90 days after study vaccination; the subject must also have a negative serum or urine pregnancy test within 14 days prior to study vaccination (if screening and study vaccination do not occur on the same day) and on the day of study vaccination prior to randomization
* Sexually active males, unless surgically sterile, must use an effective method of birth control (condom or abstinence) and must agree to continue using such precautions for at least 30 days after study vaccination
* Available by telephone
* Written informed consent (and HIPAA authorization if applicable) obtained from the subject
* Ability to understand and comply with the requirements of the protocol, as judged by the investigator
* Ability to complete follow-up period of 180 days after study vaccination as required by the protocol

Exclusion Criteria:

* History of hypersensitivity of any component of the vaccine, including egg or egg protein
* History of hypersensitivity to gentamicin
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (e.g., asthma), chronic metabolic diseases (e.g., diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (>100.0°F oral or equivalent) and/or clinically significant respiratory illness (e.g., cough or sore throat) within the 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including HIV infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome
* Household contact who is severely immunocompromised (e.g., hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual requires care in a protective environment); subject should additionally avoid close contact with severely immunocompromised individuals for at least 21 days after study vaccination
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 180 days after study vaccination (use of licensed agents for indications not listed in the package insert is permitted)
* Expected receipt of anti-pyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after study vaccination Note: A daily dose of up to 81 mg of aspirin for prophylactic use is not considered a contraindication to enrollment.
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after study vaccination
* Nursing mother
* Employee of the research center, any individual involved with the conduct of the study, or any family member of such individuals
* Any condition (e.g., chronic cough, allergic rhinitis) that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2006-06; Study Completion 2006-12

PRIMARY OUTCOMES:
The primary endpoint of this study is fever (Study Days 0-7), defined as oral temperature of at least 101°F.

SECONDARY OUTCOMES:
Secondary endpoints of the study include other reported REs and AEs that occur within 7 days after vaccination (Study Days 0-7) and all REs and AEs that occur within 14 days after vaccination (Study Days 0-14).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Allende, M.D., Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Radiant Research, Daytona Beach, Daytona Beach, Florida
  - Radiant Research, Portland, Oregon
  - Heathcare Discoveries, Inc., San Antonio, Texas